CLINICAL TRIAL: NCT04073173
Title: Stress Assessment in Preterm Infants With Respiratory Distress Syndrome Treated or Not With an Analgesic Drug During the Traditional or the Less Invasive Method of Surfactant Therapy.
Brief Title: Stress Assessment With and Without Analgesia During Surfactant Therapy in Preterm Infants.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Virgilio Paolo Carnielli (Other)
Collaborators: Fondazione Cassa di Risparmio di Verona Vicenza Belluno e Ancona (Unknown); Istituto di Ricerca Pediatrica Città della Speranza (Unknown)
Responsible Party: Sponsor-Investigator, Virgilio Paolo Carnielli, Director of Neonatology, Ospedali Riuniti Ancona
Organization: Ospedali Riuniti Ancona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: StrAAS; 2020-004269-38 (EudraCT Number)
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Distress Syndrome in Premature Infants
Keywords: RDS; Preterm Infants; Surfactant; LISA; INSURE; Analgesia; Stress
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Agnosia | interventions — Insure Cement; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and data analyst will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LISA-analgesic (Experimental): Less Invasive Surfactant Administration (LISA) with remifentanil (0.5-2 micrograms/kg/dose) as the analgesic drug.
  Interventions: Procedure: LISA; Drug: Analgesic, Opioid
- LISA-no analgesic (Experimental): Less Invasive Surfactant Administration (LISA) without an analgesic drug.
  Interventions: Procedure: LISA
- INSURE-analgesic (Experimental): INtubation-SURfactant-Extubation (INSURE) with remifentanil (0.5-2 micrograms/kg/dose) as the analgesic drug.
  Interventions: Procedure: INSURE; Drug: Analgesic, Opioid
- INSURE-no analgesic (Experimental): INSURE without an analgesic drug.
  Interventions: Procedure: INSURE

INTERVENTIONS:
Procedure: INSURE — Patients will be intubated by endotracheal tube, exogenous surfactant (Poractant alfa) will be administered and then they will be extubated.
  Arms: INSURE-analgesic; INSURE-no analgesic
Procedure: LISA — Surfactant (Poractant alfa) will be directly delivered into the lungs via a fine bore catheter inserted into the trachea and then patients will be extubated.
  Arms: LISA-analgesic; LISA-no analgesic
Drug: Analgesic, Opioid — Remifentanil (0.5-2 micrograms/kg/dose)
  Arms: INSURE-analgesic; LISA-analgesic

SUMMARY:
This study will compare stress, changes in oxygenation and oxidative damage in preterm infants with respiratory distress syndrome (RDS) randomized to receive or not remifentanil as an analgesic drug during the administration of porcine surfactant (poractant alfa, Curosurf®) through the traditional (INSURE) or the less invasive (LISA) method.

DETAILED DESCRIPTION:
At present, LISA and INSURE are both used for surfactant therapy in infants as comparable methods. However, a clear policy of using analgesics during surfactant therapy is still lacking: some neonatologists use analgesics to reduce stress and pain scores, whereas others do not approve their use due to interference with spontaneous breathing.

In this open-label, randomized, phase 4 clinical trial, infants admitted to our neonatal intensive unit care (NICU) will be evaluated according to the selection criteria and then randomized to receive or not remifentanil as an analgesic drug during the administration of porcine surfactant (poractant alfa, Curosurf®) via the INSURE or LISA method: Group-1) LISA-analgesic; Group 2) LISA-no analgesic; Group-3) INSURE-analgesic; Group-4) INSURE-no analgesic. Study patients will be stratified by gestational age at birth: Block A) 23.0-27.6 weeks of gestation; Block B) 28.0-31.6 weeks of gestation.

Early caffeine administration will be provided according to our NICU guidelines shortly after birth. Infants with adequate respiratory drive will be stabilized on nasal continuous positive airway pressure (CPAP; 4-8 cm of water) right after birth. Oxygen saturation targets will be 90-94%; moderate degrees of hypercarbia (PaCO2 < 60 mmHg, provided arterial pH >7.22) will be tolerated. Conditions mimicking respiratory distress syndrome (RDS; i.e. sepsis, air leaks, aspiration pneumonia, congenital heart disease) will be ruled out. RDS diagnosis will be clinical according to the European Guidelines. Nasal CPAP, bi-level CPAP or nasal intermittent positive pressure ventilation (synchronized or not) will be used at the discretion of the attending physician to stabilize the patients. Intubation criteria according to our NICU guidelines will be:

1. severe acidosis (defined as arterial pH<7.20 with a partial pressure of carbon dioxide (PaCO2) > 55 mmHg and partial pressure of oxygen (PaO2) < 50 mmHg) with a fraction of inspired oxygen (FiO2) > 0.50;
2. severe apnoea.

Enrolled infants will be evaluated from birth to day 7 of the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth between 168 and 223 days,
* respiratory distress syndrome (diagnosed on the basis of clinical and/or radiological grounds) with a fraction of inspired oxygen ≥0.30 (for infants born ≤26 weeks' gestational age) or ≥0.40 (for infants born >26 weeks' gestational age) to achieve a peripheral oxygen saturation of 90-94% within 24 hours of life and good respiratory drive,
* written informed consent.

Exclusion Criteria:

* major malformations,
* late admission (after 24 hours of life),
* intubation in the delivery room,
* severe birth asphyxia,
* prolonged rupture of membranes,
* air leaks,
* no informed consent.

Ages: 168 Days to 223 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Cortisol concentrations | At 1, 3, 6 12, 24 hours after surfactant administration and then daily in the first week at the same time of the day (to avoid circadian variations).
  Cortisol concentrations will be assessed in saliva, as salivary cortisol levels have been shown to be useful surrogate markers for plasma cortisol levels in neonates. Saliva samples will be collected using an absorbent swab stick, centrifuged at 4000 rpm for 10 minutes and kept at -80°C until assayed (minimum sample volume 25 µl). Enzyme immunoassay (ELISA kit) will be used. Basal samples will be obtained at the hospital admission and right before surfactant.

SECONDARY OUTCOMES:
Galvanic Skin Responses | At 1, 3, 6 12, 24 hours after surfactant administration and then daily in the first week at the same time of the day (to avoid circadian variations).
  An instrumental stress-test device measuring galvanic skin conductance will be used (Pain Monitor, Med-Storm, Norway): three electrodes will be attached to the infant's foot (sole and sides of the ankle); skin conductance is measured in micro Siemens (µS).
Heart rate | 6 hours before and after surfactant therapy will be analyzed.
  Cardiac monitoring will assess heart rate. Traces will be saved onto a computer with a sampling frequency of 1 Hertz. Average heart rate, periods of tachycardia (>160 bpm for ≥5 seconds) and bradycardia (<100 bpm for ≥5 seconds) will be recorded. These parameters may be correlated with stress and hemodynamic instability during the procedures.
Brain oxygenation | From the hospital admission to day 7 of the hospital stay.
  Brain oxygenation will be assessed by near-infrared spectroscopy (NIRS).
Oxygen saturation (SpO2) | From the hospital admission to day 7 of the hospital stay.
  High precision oxygenation assessment will be attained by high frequency (1 Hz) sampling of SpO2 data from the cardio monitor to a computer, possibly by using multiple pulse oximeters in the same patient.
Markers of oxidative stress | At the hospital admission and at 6 and 12 hours after surfactant therapy.
  8-isoprostane and nitrites/nitrates will be dosed on urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: Virgilio Carnielli, MD, PHD, Study Director — Azienda Ospedaliero-Universitaria Ospedali Riuniti di Ancona; Clementina Rondina, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Ospedali Riuniti di Ancona

REFERENCES:
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GH, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2016 Update. Neonatology. 2017;111(2):107-125. doi: 10.1159/000448985. Epub 2016 Sep 21. PMID 27649091
- [Background] Okamura H, Kinoshita M, Saitsu H, Kanda H, Iwata S, Maeno Y, Matsuishi T, Iwata O. Noninvasive surrogate markers for plasma cortisol in newborn infants: utility of urine and saliva samples and caution for venipuncture blood samples. J Clin Endocrinol Metab. 2014 Oct;99(10):E2020-4. doi: 10.1210/jc.2014-2009. Epub 2014 Jul 31. PMID 25078034
- [Background] Lago P, Benini F, Agosto C, Zacchello F. Randomised controlled trial of low dose fentanyl infusion in preterm infants with hyaline membrane disease. Arch Dis Child Fetal Neonatal Ed. 1998 Nov;79(3):F194-7. doi: 10.1136/fn.79.3.f194. PMID 10194990
- [Background] Guinsburg R, Kopelman BI, Anand KJ, de Almeida MF, Peres Cde A, Miyoshi MH. Physiological, hormonal, and behavioral responses to a single fentanyl dose in intubated and ventilated preterm neonates. J Pediatr. 1998 Jun;132(6):954-9. doi: 10.1016/s0022-3476(98)70390-7. PMID 9627585
- [Background] Guinsburg R, Kopelman BI, de Almeida MF, Miyoshi MH. [Pain in intubated and ventilated preterm neonate: multidimensional assessment and response to fentanyl analgesia]. J Pediatr (Rio J). 1994 Mar-Apr;70(2):82-90. doi: 10.2223/jped.727. Portuguese. PMID 14688879
- [Background] Badiee Z, Vakiliamini M, Mohammadizadeh M. Remifentanil for endotracheal intubation in premature infants: A randomized controlled trial. J Res Pharm Pract. 2013 Apr;2(2):75-82. doi: 10.4103/2279-042X.117387. PMID 24991608